CLINICAL TRIAL: NCT04364451
Title: Correlation of Polymorphisms of Lipoprotein Lipase (LpL) and Apolipoprotein E (Apo E) With Lipid Profile of Children With Acute Lymphoblastic Leukaemia During Therapy With L - Asparaginase
Brief Title: Correlation of Polymorphisms of Lipoprotein Lipase (LpL) and Apolipoprotein E (Apo E) With Lipid Profile of Children With Acute Lymphoblastic Eukaemia During Therapy With L - Asparaginase.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Maria Ioannidou, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: 6225/28-05-2019
Record Dates: First submitted 2020-04-10; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; Children and Adolescents; Polymorphisms of LpL and apoE; Lipid profile; Asparaginase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Apolipoproteins E; Asparaginase

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected and placed in a 4ml tube without anticoagulants. The tube will be centrifuged and the blood's serum will be isolated in order to examine the biochemical parameters of the study with the cooperation of the Biochemistry Lab of University Hospital AHEPA. Furthermore, 2ml of whole blood will be collected in a tube containing Ethylenediaminetetraacetic acid (EDTA) as the anticoagulant for use in molecular techniques. The whole blood and the serum will be stored in a temperature of -80 degree Celsius.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Correlation of Polymorphisms of Lipoprotein Lipase (LpL) and Apolipoprotein E (Apo E) With Lipid Profile of Children With Acute Lymphoblastic Leukaemia During Therapy With L - Asparaginase — Children that meet all the inclusion criteria for this study will be examined and undergo treatment with asparaginase (Experimental group) and will be compared to the corresponding teams of healthy children and children that have ailed and are off chemotherapy for at least 6 months (Control group).

SUMMARY:
Haematological malignancies constitute the most common neoplastic disease in child population, with acute leukemia occupying the number one spot with a percentage of 32.8%. In children, leukaemia is primarily encountered in its acute form (97%) and in the majority of the cases it is presented as Acute Lymphoblastic Leukaemia - ALL (80%). Acute Non-Lymphoblastic Leukemia - ANLL is encountered less frequently (17%) and it includes Acute Myelogenous Leukaemia - AML (15%) and some other rare forms (2%), while the remainder 3% corresponds to chronic leukaemia.

L-Asparaginase (L-ASP) is a fundamental component during the loading phase with regards to achieving remission of the disease and, likewise, during the maintenance phase with the intention of establishing that remission in both children and adults suffering from ALL. The cytotoxic effect of the exogenous administration of Asparaginase is caused by the depletion of the reserve of asparagine in the blood. Asparaginase (ASP) acts as a catalyst for the hydrolysis of asparagine to aspartic acid and ammonia. Asparagine is vital for protein and cell synthesis and, therefore, for their survival. The normal cells of the human body have the ability to produce asparagine from aspartic acid, with the assistance of the enzyme asparagine synthetase. However, the neoplastic cells either lack the enzyme completely or contain minute amounts of it resulting in their inability to synthesize asparagine de novo. The survival of these cells and their ability to synthesize proteins depends entirely on receiving asparagine from the blood. Thus, the administration of ASP leads to the inhibition of DNA, RNA and protein synthesis which, in turn, results in the apoptosis of these cells.

Despite L-ASP's paramount importance in the chemotherapy treatment of leukaemia, it is responsible for a plethora of toxic adverse effects that sometimes even require the termination of its administration. A critical adverse event of ASP is a disorder in the metabolism of lipids. Specifically, it appears that the activation of the endogenous pathway that produces triglycerides through hepatic synthesis leads to hypertriglyceridaemia. The liver is capable of synthesizing VLDL (Very Low Density Lipoproteins) that are rich in triglycerides. Utilising the effect of the enzyme Lipoprotein Lipase (LpL), located on the vascular endothelium, the triglycerides detach from the VLDL causing the latter to transform into IDL (Intermediate Density Lipoproteins) and afterwards into LDL (Low Density Lipoproteins). The triglycerides are later extracted from the blood circulatory system and stored in the adipose tissue, while the LDL particles connect with tissue receptors or macrophage receptors. The final products of the breakdown (coming from the peripheral hydrolysis of triglycerides with the help of LpL) of chylomicrons, VLDL, the remnants of lipoproteins, will eventually be removed by hepatic receptors. Apolipoprotein E (Apo-E) plays an important role in this procedure, it binds these remnants in the presence of LpL and hepatic lipase. Along the duration of the treatment with ASP, reduced LpL functionality is recorded, resulting in impaired plasma clearance of triglycerides and an increase in their levels, while L-ASP appears to cause disorders in other lipid factors, such as cholesterol, HDL and apolipoprotein A. Disorders of lipid metabolism have been found to be associated with polymorphisms of the LpL and Apo-E genes, sometimes with positive and sometimes with negative effects on the lipid profile and more likely participation in cardiovascular complications. The current study will evaluate, the lipid profile of children with ALL, the effect of L-ASP on the lipid profile of the aforementioned patients, as well as the correlation between the polymorphisms of Lipoprotein Lipase (LpL) and Apolipoprotein E (ApoE) with the values of the lipids during chemotherapy. Both the universal and national bibliography that pertain to the effect of ASP on the potency of LpL and App E and to the values of the lipids in children that suffer from ALL during chemotherapy with L-ASP is limited, while there exists no bibliographic reference correlating the genetic background to LpL and Apo E and the relation of the lipid profile. The current study will examine for the first time gene polymorphisms of LpL and Apo E in children with ALL during treatment with ASP.

DETAILED DESCRIPTION:
Introduction

Malignancies during childhood constitute the 2nd cause of death, following injuries worldwide. According to epidemiological data, 300,000 new cases of neoplasia present themselves every year in children and teenagers under 19 years of age1, 160,000 of which concern children under the age of 15. Haematological malignancies constitute the most common neoplastic disease in child population, with acute leukemia occupying the number one spot with a percentage of 32.8%, followed by central nervous system tumors with a percentage of 21% on the second spot and lymphoma with a percentage of 12% on the third spot.

Definition - Pathophysiology

Leukaemia (L) is defined as a group of perturbations characterized by uncontrolled proliferation of white blood cells, due to the bone marrow's primary divergence from normal and the its infiltration by immature undifferentiated stem cells. By definition, more than 20% of the bone marrow is infiltrated by stem cells. Leukaemia's exact pathogenic mechanism has not been clarified as of yet, it appears, however, to be the result of genetic mutation and damage to the multipotential haematopoietic ancestral cells, during one of their distinct stages of differentiation. This fact leads to clonal expansion and inhibition of differentiation. The leukaemic cell's immunophenotype reflects the level of differentiation achieved by the neoplastic clone. The leukaemic cells divide at a slower pace and require additional time to synthesize DNA compared to normal haematopoietic cells causing anaemia, thrombocytopenia and neutropenia. At the time of the diagnosis, the leukaemic cells could have, not only replaced the normal cells of the marrow but also expanded into extra-medullary areas.

The various types of leukaemia are exceptionally heterogeneous and, depending on the cells' origin, they are differentiated into lymphoblastic and non-lymphoblastic leukemias. Each one of the above mentioned subgroups can be encountered in its Acute Leukaemia (AL) or Chronic Leukaemia (CL) form. In the acute form, the immature cells of the haematopoietic tissue are dominant and the progression of the disease without any treatment leads quickly to death. In the chronic forms, the mature cells dominate the tissue and the development of the disease, generally, takes longer. In children, leukaemia is primarily encountered in its acute form (97%) and in the majority of the cases it is presented as Acute Lymphoblastic Leukaemia (ALL, 80%). Acute Non-Lymphoblastic Leukaemia - ANLL is encountered less frequently (17%) and it includes Acute Myelogenous Leukaemia - AML (15%) and some other rare forms (2%), while the remainder 3% corresponds to chronic leukaemia. AL occurs more often between the ages of 2 and 6 years old while the incidence is higher in boys compared to girls (1:1.3). 2.5% - 5% of children's ALL and 6% - 14% of children's AML is encountered in infants under 1 year old. The characteristic type of ALL is the B-cell ALL, which is additionally the most common in children (85%) compared to the T-cell ALL (15%) which is accompanied by masses in the lymph nodes of the mediastinum amongst other areas.

Epidemiology

In the United States of America (USA) and most of the countries of Western Europe, the frequency of leukaemia in children is 3.5 - 4.0 cases per 100,000 childhood population yearly and it is ranked as the 20th cause of death among malignancies of all ages. It is deduced from large-scale cohort studies that the incidence of childhood cancer in developed countries is rising 1% every year. The prevalence of ALL in children was detected for the first time in the 1930s in the United Kingdom (UK) and the USA. In the USA, ALL appeared first in children of European descent, and afterwards, in children of African descent in the 1960s. The frequency of ALL is lower in developing and underdeveloped countries, a fact that hints at a possible correlation between industrialization and leukaemogenesis.

Asparaginase (ASP)

The chemotherapy combination treatments used today to treat ALL have improved significantly the long-term course of the disease with the overall five-year-survival rate exceeding 80%, while the respective ratio in the 1960s was under 30%. One of the main reasons that contributed to this development is the intensive, extended and higher dosed administration of Asparaginase. L-Asparaginase (L-ASP) is a fundamental component during the loading dose with regards to achieving remission of the disease and, likewise, during the maintenance dose with the intention of establishing that remission in both children and adults suffering from ALL. The cytotoxic effect of the exogenous administration of asparaginase is caused by the depletion of the reserve of asparagine in the blood. Asparaginase acts as a catalyst for the hydrolysis of asparagine to aspartic acid and ammonia. Asparagine is vital for protein and cell synthesis and, therefore, for their survival. The normal cells of the human body have the ability to produce asparagine from aspartic acid, with the assistance of the enzyme asparagine synthetase. However, the neoplastic cells either lack the enzyme completely or contain minute amounts of it resulting in their inability to synthesize asparagine de novo. The survival of these cells and their ability to synthesize proteins depends entirely on receiving asparagine from the blood. Thus, the administration of asparaginase leads to the inhibition of DNA, RNA and protein synthesis which, in turn, results in the apoptosis of these cells. The low levels of asparagine only affect the survivability of the cancer cells, leaving the healthy cells undisturbed.

The ability of L-ASP to suppress the proliferation of the leukaemic cells was first observed in clinical studies during the 1970s, and from that moment on it has remained the cornerstone of childhood ALL treatment. The natural forms of the enzyme, produced by the bacteria Erwinia chrysanthemi and Escherichia coli (E.Coli), are being used for treatment, much like L-ASP's product created from the conjugation of E. Coli. with polyethylene glycol (Pegylated-Asparaginase, PEG-ASP) with prolonged half-life of 5.5 days instead of the 26 hour half-life of the natural forms. Chemotherapy protocols for ALL recommend a dosage of 1,000 - 2,500 IU/m2 of PEG-ASP and 5,000 - 12,000 IU/m2 of the natural form.

Adverse Reactions of Asparaginase

Despite L-ASP's paramount importance in the chemotherapy treatment of leukaemia, it is responsible for a plethora of toxic adverse effects that sometimes even require the termination of its administration. Studies have shown that the omission of administration of doses due to the emergence of toxic adverse effects in previous administrations is linked to poor prognoses in children with ALL. The most common adverse effects are hypersensitivity reactions, as studies indicate their rate occurrence is as high as 75%. The ASP that is being utilized is a large molecule of bacterial origin (mainly E. Coli) and thus is able to induce an immune response which grows more intense after repeated exposure and, mainly, after a delay of the drug administration. Aside from the clinical hypersensitivity reactions that signal an immediate response from the attending medical staff, there also exist subclinical reactions that can lead to a decrease in the potency of the drug that is difficult to detect in order to act swiftly. Pancreatitis is reported at a rate as high as 18% of the patients with ALL during treatment with ASP. The pathogenic mechanism is not yet known, however it appears that the fault lies with the decrease of protein synthesis from organs with significant protein turnover, like the pancreas. Moreover, it is considered that this mechanism is also responsible for the hepatotoxicity detected during treatment with asparaginase. Additionally, the ASP induced decrease in protein synthesis is involved in the processes of coagulation and fibrinolysis which in turn leads to thrombotic episodes of the central nervous system and deep vein thrombosis of the extremities. Other adverse reactions are hyperglycaemia, as a result of decreased insulin production and myelosuppression, mainly due to enhancing the suppression effect of the other chemotherapy drugs. Furthermore, there have been reports of incidents of encephalopathy during therapy with ASP that could be related with the elevated levels of ammonia that result from the breakdown of ASP.

A critical adverse event of ASP that could result in additional complications if it is not promptly identified is a disorder in the metabolism of lipids. Specifically, it appears that the activation of the endogenous pathway that produces triglycerides through hepatic synthesis leads to hypertriglyceridaemia. Some studies indicate that the rate of high values of triglycerides is 67% 8 - 14 days after administering the medicine. The liver is capable of synthesizing VLDL (Very Low Density Lipoproteins) that are rich in triglycerides. Utilizing the effect of the enzyme Lipoprotein Lipase (LpL), located on the vascular endothelium, the triglycerides detach from the VLDL causing the latter to transform into IDL (Intermediate Density Lipoproteins) and afterwards into LDL (Low Density Lipoproteins). The triglycerides are later extracted from the blood circulatory system and stored in the adipose tissue, while the LDL particles connect with tissue receptors or macrophage receptors. The final products of the breakdown (coming from the peripheral hydrolysis of triglycerides with the help of LpL) of chylomicrons, VLDL, the remnants of lipoproteins, will eventually be removed by hepatic receptors. Apolipoprotein E (apo-E) plays an important role in this procedure, it binds these remnants in the presence of LpL and hepatic lipase.

Lipoprotein Lipase (LpL)

The LpL gene is located on the chromosome 8p22 and is comprised of 10 exons. There have been recorded roughly 100 mutations, with 3 of them being the most common, 2 of which are connected with reduced functionality of LpL and increased cardiovascular risk. The mutation known as polymorphism N291S is present in 2-5% of the general population and its existence is associated with decreased functionality of LpL and an imbalance in the VLDL metabolism [increase of triglycerides, decrease of HDL (High Density Lipoproteins)]. In addition, it appears that the effect of this mutation is amplified by the coexistence of other genetic factors (familial hypercholesterolaemia, apolipoprotein E2/E2). The second mutation, known as polymorphism D9N, is related to increased risk of atherosclerosis, even if the mutation causes a light decrease in the functionality of LpL. As of late, it was observed that the combination of small nucleotide polymorphisms (SNP) on the genes of Apo E and of LpL denominate a high-risk group for cardiovascular disease. Lastly, the third mutation, encountered in the 20% of the general population, polymorphism S447X is linked with slightly elevated HDL levels and low levels of triglycerides and thus has a positive impact on the lipid profile.

Along the duration of the treatment with ASP, reduced LpL functionality is recorded, likely caused by the altogether reduced protein synthesis from the liver, as is apparent from the decreased concentrations of other proteins, such as albumin and fibrinogen. Studies have demonstrated, in particular, that the suppression of the LpL's effects is connected with an increase in the ratio of ApoCIII/ApoCII, where ApoCII is an essential cofactor of LpL and it promotes the hydrolysis of triglycerides and ApoCIII acts as an inhibitor of LpL while simultaneously appears to be able to regulate the levels of triglycerides in the serum independently from LpL. Hence, a problem is created in the triglyceride cleansing from the plasma as their levels rise. Another suggested mechanism for the high levels of triglycerides during treatment with asparaginase is the increase in VLDL synthesis, which is also reflected in the high apolipoprotein ApoB100 concentration, a component of VLDL.

Apolipoprotein E (Apo E)

The gene of Apo E is situated on chromosome 19 and it is comprised of 4 exons. Apolipoprotein E (Apo E) is one of the structural components included in lipoproteins, which are rich in triglycerides, and it plays an important role in the hepatic protein intake. Apolipoprotein E (Apo E) has 3 alleles ε2, ε3, ε4 [APOE-ε2 (cys112, cys158), APOE-ε3 (cys112, arg158) and APOE-ε4 (arg112, arg158)]. ε3 is the most common in the general population and it contains cysteine at position 112 and arginine at position 158. ε4 differs from ε3 at position 112, where instead of it substitutes the cysteine for arginine55. The isomorph ε2 has a weaker connection with the lipoprotein receptors of the liver which results in the accumulation of remnants from chylomicrons and VLDLs.

ApoE4 attaches to the lipoprotein receptors in the liver in vitro having the same affinity as ApoE3, however the effect of ApoE4 in the cleansing of lipoproteins rich in triglycerides in vivo is undefined as of yet. The ε2 allele is connected with higher triglyceride levels after fasting, while the ε4 allele is connected with hypercholesterolaemia and high LDL cholesterol. The individuals with the genotype E3/E4 display slower cleansing of lipoproteins rich in triglycerides in comparison with individuals with the genotype E3/E3. The ε4 allele looks to be associated with an affected triglyceride metabolism. The individuals with the ε2 allele have lower cholesterol levels compared to the individuals with ε3 and ε4 alleles. Studies indicate, further, that individuals with genotype E2/E4 have higher triglyceride levels after fasting in relation to the individuals with genotype E3/E3.

Alterations in the ApoE gene lead to changes in the amino acids of the coded protein, which results in a modified structure of the normal protein. The latter results in a slower cleansing of lipoproteins rich in triglycerides. In one study, it was revealed that there was a higher prevalence of the phenotype E4/E3 in patients with hypertriglyceridaemia compared to patients with normal triglyceride levels. Additionally, no significant statistical difference was observed between triglyceride levels and the phenotypes of ApoE after treatment with asparaginase.

Asparaginase and Lipid Profile

With regard to the effect of asparaginase on cholesterol levels, the studies do not allow to reach any reliable conclusion, as some studies found an increase in a small percentage of the patients after administering the medicine, others indicated a significant increase, while others yet presented a small but not significant decrease. Regarding the HDL levels, studies have discovered that they are lower in children suffering from malignancies, specifically of a haematological type. Another study focusing on children with ALL, during and after treatment with ASP the HDL levels rose with a simultaneous drop Apo-A1 levels. HDL plays a crucial role in the process of reverse transfer of cholesterol from the peripheral tissue to the liver, a mechanism that imparts on HDL the properties of an anticoagulant agent. Functioning in tandem with the aforementioned properties, other parts of HDL have antioxidant, anti-inflammatory, anti-apoptotic and anticoagulant properties that contribute to safeguarding against atherogenesis. Lipoprotein Apo-A1 comprises the main structural protein for HDL. It is apparent that asparaginase as an inhibitory factor of protein synthesis could possibly modify the ratio of lipids/ proteins in favor of the first on the molecules of HDL. Low HDL and Apo-A1 levels have been noticed even in free of disease survivors of ALL after the end of treatment. This observation is of particular importance if one thinks about the danger of atheromatosis and coronary disease due to low levels of HDL.

Hypertriglyceridaemia is able to become the sole contributor to the development of acute pancreatitis. When the levels of triglycerides rise above 900 mg/dl they form chylomicrons, molecules big enough in size that they can obstruct the pancreatic capillaries leading to ischaemia and release of pancreatic lipase. The latter will reinforce the lipolysis with an increase of free fatty acids which will, in turn, allow the release of free radicals and pro-inflammatory derivatives causing, in the end, inflammation and necrosis. As seen above, asparaginase is capable of taking part in the pathogenesis of pancreatitis through two routes, an independent and a dependent upon triglycerides. Hypertriglyceridaemia could also promote a predisposition for thrombosis in patients suffering from ALL and who are under treatment with ASP, as on one hand, the medicine is connected to modifications of the fibrinolytic system, as was already mentioned, meanwhile on the other hand the increase of triglycerides causes hyper-viscosity of the blood raising the risk of thromboembolic complications. Drawing from the cases documented in the universal bibliography, it is made clear that the majority of the thromboses involves the central nervous system (CNS), while on second place are cases of deep vein thrombosis of the upper extremities.

Lastly, it is significant to add that administration of ASP to children with haematological malignancies in multiple phases of the treatment is co-administrated with corticosteroids, either prednisone or dexamethasone. It can be easily perceived that corticosteroids can synergize and intensify the adverse events, such as hyperlipidaemia, pancreatitis and thrombosis. Furthermore, asparaginase can contribute to some adverse events of the corticosteroids, such as osteonecrosis through the hyper-coagulant state that it creates. Since both of these medications are pivotal therapeutic factors, a very close and attentive monitoring of the patient's condition and emergence of adverse events is required in order to intervene if necessary.

Originality

Both the universal and national bibliography that pertain to the effect of asparaginase on the potency of LpL and Apo E and to the values of the lipids in children that suffer from ALL during chemotherapy with ASP is limited, while there exists no bibliographic reference correlating the genetic background to LpL and Apo E and the relation of the lipid profile. The current study will examine for the first time gene polymorphisms of LpL and Apo E in children with acute ALL during treatment with ASP.

Importance

In this particular study investigators will focus on researching the lipid profile of children with ALL, on the effect of ASP on the lipid profile of these patients, as well the correlation between the polymorphisms of lipoprotein lipase (LpL) and Apolipoprotein E (ApoE) with the values of lipids for the duration of the chemotherapeutic protocol. The hypothesis that is going to be tested is whether recording the genotypes of the under-study children with ALL will be able to constitute a preemptive indicative factor for the outcome of their treatment.

In this manner, vital conclusions will be extracted for the probable contribution of genotypes of children that are being administered L-ASP to the laboratory demonstration of lipid disorders during treatment, the closer supervision during the corresponding phases of treatment and the timely therapeutic intervention in order to prevent any complications.

Methodology

Study Type: Prospective case-control study The characterization epidemiologic study is in complete accord with the aim of our study, a study of the effect of ASP on the lipid profile of children and adolescents with ALL (Patient Group) as well as the correlation of the polymorphisms of LpL and ApoE with the lipid levels duration of the chemotherapeutic protocol. The existence of two additional children groups that will act as population-control (children and adolescents of the same age group that do not manifest the disease and participants of the similar ages that have manifested the disease and have completed chemotherapy as per protocol for at least 6 months prior) specialises our study type into a case-control study.

Study Site: The study will be conducted in the Paediatric and Adolescent Haematology - Oncology Unit of the 2nd Department of Paediatrics, Aristotle University of Thessaloniki (AUTH), at University General Hospital AHEPA.

Description of the recorded parameters

During the disease's diagnosis, the lipid profile of the patients' will be determined by measuring the following parameters: total cholesterol, triglycerides, HDL-cholesterol, LDL-cholesterol, apolipoprotein A1, apolipoprotein B100, lipoprotein α [Lp(α)], glucose, Serum Glutamic Oxaloacetic Transaminase (SGOT), Serum Glutamic Pyruvic Transaminase (SGPT),Thyroid-Stimulating Hormone (TSH), Free Thyroxine (FT4), amylase, lipase. Additionally, a genetic analysis for polymorphisms of LpL and Apo E will be conducted. Similar measurements will be done to all participants of all groups.

The participants of group A will be immediately subjected to the chemotherapy protocol ALLIC BFM 2009. During the loading dose, these children will receive treatment with prednisolone for 33 consecutive days and asparaginase will be added on days 12, 15, 18, 21, 24, 27, 30, 33. During the maintenance phase the children will be subjected anew to treatment with corticosteroids, dexamethasone, and asparaginase will be added on days 8, 11, 16, 18. The lipid identity will be checked before administration of ASP on day 0 and 11 as well as after the administration of ASP and before the administration of the next dose at the loading dose, meaning days 15, 24, 33. Similarly, the lipid identity will be checked on the maintenance phase, meaning on days 8, 16, 21 as well as after the end of every phase of chemotherapy protocol in which ASP is not administered.

Moreover, an examination of LpL polymorphisms (the three most common polymorphisms p.N291S, p.D9N, p.S447X) and of Apo E polymorphisms [ε2(rs7412-T,rs429358-T), ε3(rs7412-C, rs429358-T) and ε4 (rs7412-C, rs429358-C)] will be performed after isolating the DNA from the peripheral blood and analyzing it with molecular techniques.

Participants that meet all the inclusion criteria for this study will be examined and undergo treatment with ASP (Patient group) and will be compared to the corresponding teams of healthy children and children that have ailed and are off chemotherapy for at least 6 months (Controls group).

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents newly diagnosed with acute lymphoblastic leukaemia. A complete personal and family history will be recorded for each participant from every group with particular emphasis on the presence of dyslipidaemia, early cardiovascular disease or cerebrovascular accident in the individual or in the family. A thorough clinical examination will be performed and the vital signs, blood pressure, weight (kg), height (m) and a Body/Mass Index (BMI) will be recorded and calculate.

The Exclusion criteria are the following:

* Thyroid Disorder (Abnormal thyroid function)
* Familial Hypercholesterolemia
* High Body/ Mass Index (BMI)
* Administration of corticosteroids some time during the past 2 weeks before diagnosis
* Administration of total parenteral nutrition before the diagnosis
* Administration of plasma before the diagnosis
* Changes or variation of the parameters under study before the start of treatment and the 11th day (before the start of asparagine administration).

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Prospective children and adolescents will participate, newly diagnosed with acute lymphoblastic leukaemia, which will be thoroughly tested for a precise and accurate diagnosis of acute leukaemia. Those children will create Team A (Patient Group). Furthermore, an equivalent number of children will participate, of similar ages that have been ailing from ALL and have terminated their chemotherapy for more than 6 months. These children will compose Team B (Control group).
  In addition, in the control group (Team C) children will be added of similar ages that have not ailed from ALL (Healthy control group).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The correlation of lipoprotein lipase (LpL) and apolipoprotein E (apoE) polymorphisms with lipid values during the chemotherapy protocol. | Baseline
  The genotypes of children with ALL will be recorded and it might constitute an early indicative factor concerning the treatment's outcome. Thusly, essential information will be extracted about the possible contribution of genotype of children under treatment with L-ASP to the lipid disorder as shown in the lab results, to better monitoring of each unique phase of the therapy for clinical occurrences and complication and to faster therapeutic intervention.
Assessment of the effect of asparaginase by measuring the changes induced in the lipid profile of children with acute lymphoblastic leukaemia. | Baseline and days 11, 15, 24, 33 in loading phase and days 8, 16, 21 in maintenance phase
  During the disease's diagnosis, the lipid profile of the patients' will be determined by measuring the changes of the following parameters compared to the baseline measures: cholesterol (mg/dl), triglycerides(mg/dl), HDL-cholesterol(mg/dl), LDL-cholesterol(mg/dl), apolipoprotein A1(mg/dl), apolipoprotein B100(g/L), lipoprotein α [Lp(α)](nmol/l), glucose (mg/dl), SGOT (U/I), SGPT (U/I), TSH (mU/l) FT4 (pmol/l) amylase (U/I) and lipase (U/I).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Hatzipantelis, As.Professor, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- Paediatric and Adolescent Haematology-Oncology Unit, 2nd Department of Paediatrics, Aristotle University of Thessaloniki (AUTH), University General Hospital AHEPA, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided